CLINICAL TRIAL: NCT07252323
Title: A Single-arm Phase II Clinical Study Investigating the Safety and Efficacy of Carbon Ion Radiotherapy in Patients With Hepatocellular Carcinoma Previously Treated With Transarterial Radioembolization (TARE)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2024-1588
Record Dates: First submitted 2025-11-18; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Carcinoma; Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma; Carcinoma, Hepatocellular | interventions — Heavy Ion Radiotherapy

STUDY DESIGN:
Intervention Model Description: All enrolled participants will receive carbon ion radiotherapy as a single-arm interventional treatment. Outcomes will be evaluated prospectively to assess safety and efficacy in patients with hepatocellular carcinoma previously treated with TARE.
Masking Description: This is an open-label study; no blinding will be applied to participants, investigators, or outcome assessors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Carbon Ion Radiotherapy (Experimental): Participants will receive carbon ion radiotherapy targeting residual or recurrent hepatocellular carcinoma following prior transarterial radioembolization (TARE). Treatment will be delivered using hypofractionated high-linear energy transfer radiation, with dose and fractionation individualized based on tumor size, anatomical location, and organ-at-risk constraints. The intervention aims to provide effective local tumor control while maintaining acceptable safety in patients who have limited subsequent treatment options after TARE.
  Interventions: Radiation: Carbon Ion Radiotherapy

INTERVENTIONS:
Radiation: Carbon Ion Radiotherapy — Carbon ion radiotherapy will be delivered to residual or recurrent hepatocellular carcinoma in patients previously treated with transarterial radioembolization (TARE). Treatment will be administered using hypofractionated high-linear energy transfer radiation, with dose and fractionation individualized based on tumor size, tumor location, and organ-at-risk constraints. The aim of the intervention is to achieve enhanced local tumor control while minimizing toxicity to surrounding normal tissues

SUMMARY:
This is a prospective, single-arm Phase II study designed to evaluate the safety and efficacy of carbon ion radiotherapy in patients with hepatocellular carcinoma (HCC) who demonstrate residual or recurrent disease after prior transarterial radioembolization (TARE). Carbon ion radiotherapy delivers highly conformal, high-linear energy transfer radiation, enabling dose escalation to hepatic tumors while minimizing exposure to surrounding normal tissues.

Eligible patients will receive carbon ion radiotherapy to target lesions, and clinical outcomes including objective response rate, progression-free survival, overall survival, and treatment-related toxicity will be systematically assessed. The study aims to determine whether carbon ion radiotherapy can provide effective local tumor control and acceptable safety in this population, thereby establishing evidence to guide its therapeutic role following TARE.

DETAILED DESCRIPTION:
This prospective, single-arm Phase II study evaluates the safety and efficacy of carbon ion radiotherapy in patients with hepatocellular carcinoma (HCC) who have residual or recurrent disease after prior transarterial radioembolization (TARE). Although TARE is an important locoregional treatment, some patients exhibit incomplete response or local progression and have limited subsequent therapeutic options.

Carbon ion radiotherapy provides highly conformal dose distribution and increased biological effectiveness, enabling escalation of tumoricidal doses while sparing surrounding liver tissue and adjacent gastrointestinal organs. Eligible patients will undergo baseline assessments and multidisciplinary review to confirm suitability for treatment. Carbon ion radiotherapy will be delivered using hypofractionated regimens individualized based on tumor characteristics and organ-at-risk constraints.

Patients will be followed with scheduled imaging, laboratory tests, and toxicity assessments. Efficacy will be measured through tumor response, local control, progression-free survival, and overall survival. Safety will be evaluated according to CTCAE criteria. The study aims to determine whether carbon ion radiotherapy can serve as an effective and feasible salvage treatment for TARE-refractory or recurrent HCC.

ELIGIBILITY:
Inclusion Criteria:

* adult patients over the age of 19 Hepatocellular carcinoma patients confirmed imagingly or histologically Patients who have a residual lesion in the TARE-treated area or have a recurrence or progressive lesion in the TARE-treated area or nearby liver and are deemed to need additional treatment when evaluating the response for more than 6 months Child-Pugh Class A (Child-Pugh score 5-6), B (CP score 7) Patients who fall within the range of lesions that can afford the baryon treatment intended in this study Patients who have minimal availability of liver excluded from treatment in terms of preservation of liver function proper liver function Patients with AST/ALT less than 5 times the upper limit of normal If you don't have blood clotting disorder ECOG performance status 2 or lower Patients who are not pregnant or who are undergoing appropriate contraception for women of childbearing age No other underlying conditions that seriously affect survival Patients who have listened to and agreed to a documented explanation and a statement of consent

Exclusion Criteria:

* If you've had external radiotherapy in your liver Patients with unresolved infections at that point Patients who have a current or other history of advanced carcinoma within 5 years a patient who underwent a liver transplant If baryon treatment is inappropriate or dangerous under the judgment of a radiologic oncologist

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-11-12 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to 6 months after completion of carbon ion radiotherapy
  Objective response rate is defined as the proportion of patients achieving complete response (CR) or partial response (PR) according to mRECIST criteria. Tumor response will be assessed through scheduled imaging studies within 6 months after carbon ion radiotherapy.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up to 3 years after initiation of carbon ion radiotherapy
  PFS is defined as the time from the start of carbon ion radiotherapy to the first documented disease progression or death from any cause, or to the date of last follow-up.
Overall Survival (OS) | Up to 3 years after initiation of carbon ion radiotherapy
  OS is defined as the time from the start of carbon ion radiotherapy to death from any cause, or to the last follow-up date for censored patients.
Time to overall tumor progression (TTP) | Up to 3 years after initiation of carbon ion radiotherapy
  TTP is defined as the time from the start of carbon ion radiotherapy to progression of any target or non-target lesion, or the appearance of new intrahepatic or extrahepatic lesions.
Time to local progression | Up to 3 years after initiation of carbon ion radiotherapy
  Time to local progression is defined as the interval from the start of carbon ion radiotherapy to radiologic progression within the treated liver area.
Treatment-related toxicity | From treatment initiation through 30 days post-treatment, or until the next alternative therapy
  Toxicity will be evaluated and graded according to CTCAE version 5.0. Toxicity follow-up continues from treatment initiation until confirmation of study completion or until the earliest start of subsequent therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided